CLINICAL TRIAL: NCT01113957
Title: A Phase 2 Randomized Clinical Trial of ABT-888 in Combination With Temozolomide Versus Pegylated Liposomal Doxorubicin Alone in Subjects With Recurrent High Grade Serous Ovarian Cancer
Brief Title: A Trial of ABT-888 in Combination With Temozolomide Versus Pegylated Liposomal Doxorubicin Alone in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-757; 2009-015082-31 (EudraCT Number)
Record Dates: First submitted 2010-02-26; First posted 2010-04-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2014-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — veliparib; liposomal doxorubicin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): ABT-888 in combination with temozolomide
  Interventions: Drug: ABT-888; Drug: temozolomide
- Arm B (Active Comparator): pegylated liposomal doxorubicin alone
  Interventions: Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: ABT-888 — Arm-A subjects will be given ABT-888 on Days 1 -7 every 28 days orally
  Other Names: ABT-888, veliparib
  Arms: Arm A
Drug: pegylated liposomal doxorubicin — Arm B subjects randomized to pegylated liposomal doxorubicin on Day 1, every 28 days intravenously.
  Other Names: doxil/caelyx
  Arms: Arm B
Drug: temozolomide — Arm A subjects will be given temozolomide on days 1-5 every 28 days orally with ABT-888
  Other Names: temozolomide, temodar/temodal
  Arms: Arm A

SUMMARY:
The purpose of this study is to determine the objective response rate of ABT-888 when given in combination with temozolomide versus pegylated liposomal doxorubicin (PLD) alone in subjects with recurrent high grade serous ovarian cancer.

DETAILED DESCRIPTION:
Safety assessments and tolerability will be assessed through electrocardiograms (ECG). clinical laboratory tests, vital signs, Adverse Event assessments, and physical exams. Baseline radiographic tumor assessments, including CT scans of the chest, abdomen and pelvis will be obtained. Radiologic assessments and CA-125 measurements will also be performed every 8 weeks during dosing and following completion of dosing until disease progression. Study visits will be conducted weekly for the first 2 cycles and on Day 1 of each subsequent cycle, at the Final Visit and 30 day Follow-up Visit. Study visits will include physical examination, complete blood count (CBC) and chemistries. A urinalysis tests will be performed at Screening and Final Visit. An ECG will be performed at Screening, Cycle 1 Day 1 and at the Final Study Visit. A left ventricular ejection fraction (LVEF) will be measured by Echocardiogram or Multiple Gated Acquisition (MUGA) scan on all subjects at Screening. Subjects randomized to the PLD arm will have an echocardiogram or MUGA performed at the Final Study Visit and at the discretion of the Investigator throughout the study. Adverse events will be assessed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histologically (or cytologically) confirmed recurrent high grade serous ovarian, fallopian tube, or primary peritoneal cancer.
* Subjects must have had at least 1 platinum containing chemotherapy regimen and no more than a total of 3 DNA damaging or cytotoxic regimens in the last 5 years. Less than a full dose of a DNA damaging agent, possibly due to reasons such as toxicity or documented allergic reaction are allowed. Previous treatments with biologics (including catumaxomab, tigatuzumab, abagovomab, and bevacizumab), vaccines, immunostimulants, hormonal agents, and signal transduction inhibitors (e.g., pazopanib, sorafenib, sunitinib, temsirolimus) are allowed and are not counted towards the limit of 3.
* Subjects who are resistant to platinum-based therapy; or sensitive to but are unable to tolerate platinum-based therapy (i.e., deemed toxic or have a documented platinum allergy). Subjects must have at least a > 3 month treatment free interval from the last dose of platinum based therapy.
* Subject must be eligible for PLD treatment.
* Subject has either:

  * Measurable disease, defined as at least 1 unidimensionally measurable lesion on a computed tomography (CT) scan as defined by response evaluation criteria in solid tumors (RECIST) version 1.1 OR
  * Non-measurable disease with an elevation of serum CA-125 level by Gynecologic Cancer Intergroup (GCIG) criteria (baseline sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment).
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* Subject must have adequate hematologic, renal and hepatic function as follows:

  * Bone Marrow: Absolute neutrophil count (ANC ≥ 1,500/mm3 (1.5 x 109/L); Platelets ≥ 100,000/mm3 (100 x 109/L); Hemoglobin ≥ 9.5 g/dL (1.4 mmol/L);
  * Renal function: Serum creatinine ≤ 1.5 x upper normal limit of institution's normal range OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal;
  * Hepatic function: Aspartate aminotransferase (AST) and/or alanine transaminase (ALT) ≤ 2.5 x the upper normal limit of institution's normal range. For subjects with liver metastases, AST and/or ALT < 5 x the upper normal limit of institution's normal range; Bilirubin ≤ 1.5 x the upper normal limit of institution's normal range;
  * Partial thromboplastin time (PTT) must be ≤ 1.5 x the upper normal limit of institution's normal range and international normalized ratio (INR) < 1.5. Subjects on anticoagulant (such as Coumadin) are allowed on study and will have PTT and INR as determined by the Investigator
* Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and for 90 days following completion of therapy. Women of childbearing potential must have a negative serum pregnancy test within 21 days prior to initiation of treatment and a negative urine pregnancy test on Cycle 1 Day 1. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

* Subject has previously received a poly-ADP-ribose)-polymerase (PARP) inhibitor except a single dose from Cancer Therapy Evaluation Program (CTEP) Phase 0 (A06-161) study.
* Subjects who have a history of hypersensitivity reactions to a conventional formulation of doxorubicin hydrocloride (HCL) or the components of PLD.
* The subject has received an anticancer agents or an investigational agent within 28 days prior to study drug administration. Subjects who have not recovered to within one grade level (not to exceed grade 2) of their baseline following a significant adverse event or toxicity attributed to previous anticancer treatment are excluded.
* Subject has undergone major surgery within the previous 28 days prior to study drug administration.
* Subjects with prior radiotherapy to any portion of the abdominal cavity and pelvis, unless for the treatment of ovarian, primary peritoneal or fallopian tube cancer. Subject must have completed radiation at least 28 days prior to study drug administration and have measurable disease outside the radiation field or documented progression of lesions within a previously radiated field.
* Subjects with a known history of brain metastases.
* Clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * Active uncontrolled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
  * Any medical condition, which is in the opinion of the Study Investigator, places the subject at an unacceptably high risk for toxicities
* Subject is pregnant or lactating.
* Subjects who requires parenteral nutrition, or tube feeding or has evidence of partial bowel obstruction or perforation.
* The subject has had another active malignancy within the past five years except for any cancer in situ considered cured or non-melanoma carcinoma of the skin. Questions regarding the inclusion of individual subject should be directed to the Abbott Medical Monitor.
* Subject has previously received a poly-ADP-ribose)-polymerase (PARP) inhibitor except a single dose from Cancer Therapy Evaluation Program (CTEP) Phase 0 (A06-161) study. - Subjects who have a history of hypersensitivity reactions to a conventional formulation of doxorubicin hydrocloride (HCL) or the components of PLD.
* The subject has received an anticancer agents or an investigational agent within 28 days prior to study drug administration. Subjects who have not recovered to within one grade level (not to exceed grade 2) of their baseline following a significant adverse event or toxicity attributed to previous anticancer treatment are excluded.
* Subject has undergone major surgery within the previous 28 days prior to study drug administration.
* Subjects with prior radiotherapy to any portion of the abdominal cavity and pelvis, unless for the treatment of ovarian, primary peritoneal or fallopian tube cancer. Subject must have completed radiation at least 28 days prior to study drug administration and have measurable disease outside the radiation field or documented progression of lesions within a previously radiated field.
* Subjects with a known history of brain metastases.
* Clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * Active uncontrolled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
  * Any medical condition, which is in the opinion of the Study Investigator, places the subject at an unacceptably high risk for toxicities
  * Subject is pregnant or lactating.
  * Subjects who requires parenteral nutrition, or tube feeding or has evidence of partial bowel obstruction or perforation.
* The subject has had another active malignancy within the past five years except for any cancer in situ considered cured or non-melanoma carcinoma of the skin. Questions regarding the inclusion of individual subject should be directed to the Abbott Medical Monitor.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate between the two treatment arms (ABT-888 + temozolomide versus the PLD) will be based on tumor measurements and CA-125 levels. | Screening to survival follow-up (every 3 months for 3 years)

SECONDARY OUTCOMES:
Evaluate progression free survival, time to progression, overall survival, 12-month survival rate, 6-month progression free survival rate, duration of response | Screening to survival follow-up (every 3 months for 3 years)
Safety Assessments and tolerability (i.e. ECG, clinical laboratory tests, vital signs, AE assessments, physical exams, CT scans). See section 5 for detailed information. | Screening to the 30 day follow-up visit
Evaluate Quality of Life and performance status will be done through the use of FACT-O quality of fife questionnaire, EQ5D questionnaire and ECOG performance status. | Screening to survival follow-up (every 3 months for 3 years).

CONTACTS AND LOCATIONS:
Overall Officials: Mark D McKee, MD, Study Director — AbbVie
Locations (32):
- United States (15):
  - Site Reference ID/Investigator# 25028, Duarte, California
  - Site Reference ID/Investigator# 25024, Encino, California
  - Site Reference ID/Investigator# 25034, Los Angeles, California
  - Site Reference ID/Investigator# 25037, Newport Beach, California
  - Site Reference ID/Investigator# 25030, Chicago, Illinois
  - Site Reference ID/Investigator# 27837, Park Ridge, Illinois
  - Site Reference ID/Investigator# 25039, Peoria, Illinois
  - Site Reference ID/Investigator# 25038, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 25023, New York, New York
  - Site Reference ID/Investigator# 25041, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 25029, Hilliard, Ohio
  - Site Reference ID/Investigator# 25543, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 25036, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 25042, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 25027, Houston, Texas
- Australia (6):
  - Site Reference ID/Investigator# 25128, Adelaide
  - Site Reference ID/Investigator# 25130, Bedford Park
  - Site Reference ID/Investigator# 25131, East Melbourne
  - Site Reference ID/Investigator# 25133, Nedlands
  - Site Reference ID/Investigator# 25132, Randwick
  - Site Reference ID/Investigator# 25129, Westmead
- Canada (3):
  - Site Reference ID/Investigator# 25166, Edmonton
  - Site Reference ID/Investigator# 25162, Kelowna
  - Site Reference ID/Investigator# 25165, Laval
- Site Reference ID/Investigator# 25135, Budapest, Hungary
- Israel (3):
  - Site Reference ID/Investigator# 25138, Haifa
  - Site Reference ID/Investigator# 25139, Tel Aviv
  - Site Reference ID/Investigator# 25141, Tel Litwinsky
- Site Reference ID/Investigator# 25402, Auckland, New Zealand
- Site Reference ID/Investigator# 25145, Warsaw, Poland
- United Kingdom (2):
  - Site Reference ID/Investigator# 25149, Northwood
  - Site Reference ID/Investigator# 25154, Oxford

REFERENCES:
- [Background] Elit L, Hirte H. Palliative systemic therapy for women with recurrent epithelial ovarian cancer: current options. Onco Targets Ther. 2013;6:107-18. doi: 10.2147/OTT.S30238. Epub 2013 Feb 26. PMID 23459506